CLINICAL TRIAL: NCT00993382
Title: Double Blind Placebo Controlled Dose Ranging Study of the Efficacy and Safety of Celivarone at 50, 100 or 300 mg OD With Amiodarone as Calibrator for the Prevention of ICD Interventions or Death
Brief Title: Dose Ranging Study of Celivarone With Amiodarone as Calibrator for the Prevention of Implantable Cardioverter Defibrillator (ICD) Interventions or Death
Acronym: ALPHEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DRI10936; 2008-008412-47 (EudraCT Number)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Arrhythmia Prophylaxis; Ventricular Arrhythmia
MeSH Terms: interventions — celivarone; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Celivarone 50 mg (Experimental): Celivarone, 50 mg once daily up to 10-15 days before the common study end date
  Interventions: Drug: Celivarone; Drug: Matching placebo
- Celivarone 100 mg (Experimental): Celivarone, 100 mg once daily up to 10-15 days before the common study end date
  Interventions: Drug: Celivarone; Drug: Matching placebo
- Celivarone 300 mg (Experimental): Celivarone, 300 mg once daily up to 10-15 days before the common study end date
  Interventions: Drug: Celivarone; Drug: Matching placebo
- Amiodarone (Active Comparator): Amiodarone, 600 mg once daily for 10 days (loading dose) then 200 mg once daily up to 10-15 days before the common study end date
  Interventions: Drug: Amiodarone; Drug: Matching placebo
- Placebo (Placebo Comparator): Matching placebo once daily up to 10-15 days before the common study end date
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Celivarone — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: SSR149744
  Arms: Celivarone 100 mg; Celivarone 300 mg; Celivarone 50 mg
Drug: Amiodarone — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Cordarone
  Arms: Amiodarone
Drug: Matching placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Matching placebo added to active drug if any for a total of 3 capsules per intake

SUMMARY:
The Primary objective was to assess the efficacy of Celivarone for the prevention of Implantable Cardioverter Defibrillator (ICD) interventions or death.

Secondary objectives were:

* To assess the tolerability and safety of the different dose regimens of Celivarone in the selected population.
* To document Celivarone plasma levels during the study.

DETAILED DESCRIPTION:
The study included a one week screening period, followed by a treatment period ranging between 6 and 19 months.

The treatment was to be continued until the End of Treatment visit scheduled 10-15 days prior to the common Scheduled Study End Date (SSED). The SSED was defined as about 190 days after the last patient randomization date.

The expected recruitment duration was about 14 months and thus the total duration of the study about 20 months. Visits were planned to be performed at baseline, after 5 days, after 14 days, every month for 6 months and then, every three months after 6 months until the end of the study.

ELIGIBILITY:
Inclusion criteria :

* Implantable Cardioverter Defibrillator (ICD) patients with a Left Ventricular Ejection Fraction (LVEF) of 40% or less AND one of the following criteria:

  * at least one ICD therapy for Ventricular Tachycardia (VT) OR
  * Ventricular Fibrillation (VF) in the previous month OR
  * ICD implantation in the previous month for documented VT/VF

Exclusion criteria :

* Patients of either sex aged below 21 years (or the age of legal consent of the country),
* Women of childbearing potential without adequate birth control or pregnant or breastfeeding women
* Patients with known ICD lead problem (lead dislodgement)
* ICD without the following characteristics :

  * data logging function with cumulative counting of device intervention (shocks and anti-tachycardia pacing [ATP])
  * electrogram storage capabilities
  * ventricular demand pacing.
* Recent unstable angina pectoris or myocardial infarction (< 4 weeks),
* History of torsades de pointes,
* Genetic channelopathies including congenital long QT syndrome,
* Wolff-Parkinson-White syndrome,
* Patients in unstable hemodynamic condition such as acute pulmonary edema within 12 hours prior to start of study medication; cardiogenic shock; treatment with intravenous pressor agents; patients on respirator; congestive heart failure of stage New York Heart Association (NYHA) IV within the last 4 weeks; uncorrected, hemodynamically significant primary obstructive valvular disease; hemodynamically significant obstructive cardiomyopathy; a cardiac operation or revascularization procedure within 4 weeks preceding randomization,
* Incessant sustained VT/VF (VT/VF that recurs promptly despite termination attempts) during the three days preceding randomization.
* Patients with inappropriate (not triggered by VT nor VF) shocks during the month preceding randomization.
* Clinically relevant haematologic, hepatobiliary (ALT, AST > 3 times the upper limit of normal at randomization), gastro-intestinal, renal (serum creatinine > 221 µmol/l (2.5 mg/dl) at randomization), pulmonary, endocrinologic or psychiatric disease.
* Patients treated with oral amiodarone (more than 20 tablets during the 2 months preceding randomization)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time to Ventricular Tachycardia or Ventricular Fibrillation (VT/VF) triggered ICD interventions or sudden death | up to 20 months (median follow-up of 12 months)
  The presence of VT or VF was documented by ICD interrogation leading to any ICD interventions (shocks or anti-tachycardia pacing).
  The 10 first ICD interventions for each patient were centrally and blindly adjudicated by an Adjudication Committee.

SECONDARY OUTCOMES:
Time to ICD shocks (appropriate or inappropriate) or death from any cause | up to 20 months (median follow-up of 12 months)
Time to Cardiovascular hospitalization or death | up to 20 months (median follow-up of 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Peter KOWEY, Pr, Study Chair — Steering Committee Chair Person
Locations (151):
- United States (37):
  - Investigational Site Number 840006, Huntsville, Alabama
  - Investigational Site Number 840042, Mobile, Alabama
  - Investigational Site Number 840014, Mesa, Arizona
  - Investigational Site Number 840032, Phoenix, Arizona
  - Investigational Site Number 840033, Tucson, Arizona
  - Investigational Site Number 840054, Redondo Beach, California
  - Investigational Site Number 840007, Redwood City, California
  - Investigational Site Number 840039, Colorado Springs, Colorado
  - Investigational Site Number 840002, Fort Myers, Florida
  - Investigational Site Number 840010, Orlando, Florida
  - Investigational Site Number 840005, Port Charlotte, Florida
  - Investigational Site Number 840013, St. Petersburg, Florida
  - Investigational Site Number 840043, St. Petersburg, Florida
  - Investigational Site Number 840004, Augusta, Georgia
  - Investigational Site Number 840045, Chicago, Illinois
  - Investigational Site Number 840035, Lombard, Illinois
  - Investigational Site Number 840017, Kansas City, Kansas
  - Investigational Site Number 840022, Scarborough, Maine
  - Investigational Site Number 840009, Ann Arbor, Michigan
  - Investigational Site Number 840026, Detroit, Michigan
  - Investigational Site Number 840003, Petoskey, Michigan
  - Investigational Site Number 840015, Ypsilanti, Michigan
  - Investigational Site Number 840049, Columbia, Missouri
  - Investigational Site Number 840019, Kansas City, Missouri
  - Investigational Site Number 840031, New York, New York
  - Investigational Site Number 840029, Tulsa, Oklahoma
  - Investigational Site Number 840037, Portland, Oregon
  - Investigational Site Number 840024, Camp Hill, Pennsylvania
  - Investigational Site Number 840030, Doylestown, Pennsylvania
  - Investigational Site Number 840034, Upland, Pennsylvania
  - Investigational Site Number 840020, Charleston, South Carolina
  - Investigational Site Number 840048, Rapid City, South Dakota
  - Investigational Site Number 840011, Tullahoma, Tennessee
  - Investigational Site Number 840025, Chesapeake, Virginia
  - Investigational Site Number 840012, Norfolk, Virginia
  - Investigational Site Number 840038, Richmond, Virginia
  - Investigational Site Number 840016, Spokane, Washington
- Argentina (3):
  - Investigational Site Number 032002, Ciudad Autonoma de Bs.As
  - Investigational Site Number 032003, Corrientes
  - Investigational Site Number 032004, San Miguel de Tucumán
- Australia (11):
  - Investigational Site Number 036012, Adelaide
  - Investigational Site Number 036006, Auchenflower
  - Investigational Site Number 036004, Bedford Park
  - Investigational Site Number 036014, Camperdown
  - Investigational Site Number 036013, Garran
  - Investigational Site Number 036010, Gosford
  - Investigational Site Number 036005, Herston
  - Investigational Site Number 036008, Nedlands
  - Investigational Site Number 036009, New Lambton
  - Investigational Site Number 036007, Perth
  - Investigational Site Number 036003, Woolloongabba
- Belgium (6):
  - Investigational Site Number 056005, Aalst
  - Investigational Site Number 056007, Bruges
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056002, Gilly
  - Investigational Site Number 056004, Hasselt
  - Investigational Site Number 056003, Roeselare
- Canada (9):
  - Investigational Site Number 124009, Calgary
  - Investigational Site Number 124010, Hamilton
  - Investigational Site Number 124004, London
  - Investigational Site Number 124008, Montreal
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124005, Ste-Foy
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124006, Vancouver
  - Investigational Site Number 124007, Victoria
- Investigational Site Number 152001, Santiago, Chile
- Czechia (6):
  - Investigational Site Number 203004, Brno
  - Investigational Site Number 203002, České Budějovice
  - Investigational Site Number 203005, Hradec Králové
  - Investigational Site Number 203001, Liberec
  - Investigational Site Number 203003, Olomouc
  - Investigational Site Number 203006, Prague
- Denmark (4):
  - Investigational Site Number 208002, Aarhus
  - Investigational Site Number 208004, Hellerup
  - Investigational Site Number 208005, København Ø
  - Investigational Site Number 208001, Odense C
- Finland (2):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246004, Tampere
- France (7):
  - Investigational Site Number 250004, Brest
  - Investigational Site Number 250006, Grenoble
  - Investigational Site Number 250005, Lille
  - Investigational Site Number 250002, Montpellier
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250007, Rennes
  - Investigational Site Number 250003, Vandœuvre-lès-Nancy
- Germany (5):
  - Investigational Site Number 276005, Bad Neustadt an der Saale
  - Investigational Site Number 276002, Bernau
  - Investigational Site Number 276003, Dresden
  - Investigational Site Number 276001, Frankfurt am Main
  - Investigational Site Number 276006, Hamburg
- Hungary (4):
  - Investigational Site Number 348001, Balatonfüred
  - Investigational Site Number 348004, Budapest
  - Investigational Site Number 348005, Pécs
  - Investigational Site Number 348003, Zalaegerszeg
- Israel (4):
  - Investigational Site Number 376002, Afula
  - Investigational Site Number 376003, Ashkelon
  - Investigational Site Number 376004, Haifa
  - Investigational Site Number 376001, Tel Aviv
- Italy (5):
  - Investigational Site Number 380004, Bari
  - Investigational Site Number 380008, Bergamo
  - Investigational Site Number 380002, Como
  - Investigational Site Number 380001, Florence
  - Investigational Site Number 380007, Roma
- Japan (6):
  - Investigational Site Number 392004, Meguro-Ku
  - Investigational Site Number 392005, Niigata
  - Investigational Site Number 392006, Osaka
  - Investigational Site Number 392001, Osaka Sayama-Shi
  - Investigational Site Number 392003, Shinjuku-Ku
  - Investigational Site Number 392002, Suita-Shi
- Investigational Site Number 484002, Mexico City, Mexico
- Netherlands (6):
  - Investigational Site Number 528001, Alkmaar
  - Investigational Site Number 528005, Amsterdam
  - Investigational Site Number 528002, Breda
  - Investigational Site Number 528003, Maastricht
  - Investigational Site Number 528007, Rotterdam
  - Investigational Site Number 528004, Zwolle
- Investigational Site Number 578003, Drammen, Norway
- Poland (7):
  - Investigational Site Number 616007, Bydgoszcz
  - Investigational Site Number 616011, Gdynia
  - Investigational Site Number 616006, Lodz
  - Investigational Site Number 616003, Lodz
  - Investigational Site Number 616002, Szczecin
  - Investigational Site Number 616008, Warsaw
  - Investigational Site Number 616001, Warsaw
- Portugal (3):
  - Investigational Site Number 620004, Coimbra
  - Investigational Site Number 620003, Lisbon
  - Investigational Site Number 620005, Vila Nova de Gaia
- Russia (7):
  - Investigational Site Number 643005, Moscow
  - Investigational Site Number 643003, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643008, Samara
  - Investigational Site Number 643004, Tomsk
  - Investigational Site Number 643007, Tyumen
  - Investigational Site Number 643006, Yekaterinburg
- Slovakia (2):
  - Investigational Site Number 703001, Bratislava
  - Investigational Site Number 703002, Košice
- Investigational Site Number 710002, Pretoria, South Africa
- Spain (7):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724006, Santiago de Compostela
  - Investigational Site Number 724009, Seville
  - Investigational Site Number 724007, Valencia
- Sweden (3):
  - Investigational Site Number 752002, Stockholm
  - Investigational Site Number 752003, Umeå
  - Investigational Site Number 752001, Uppsala
- Turkey (Türkiye) (3):
  - Investigational Site Number 792001, Ankara
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792002, Istanbul

REFERENCES:
- [Result] Kowey PR, Crijns HJ, Aliot EM, Capucci A, Kulakowski P, Radzik D, Roy D, Connolly SJ, Hohnloser SH; ALPHEE Study Investigators. Efficacy and safety of celivarone, with amiodarone as calibrator, in patients with an implantable cardioverter-defibrillator for prevention of implantable cardioverter-defibrillator interventions or death: the ALPHEE study. Circulation. 2011 Dec 13;124(24):2649-60. doi: 10.1161/CIRCULATIONAHA.111.072561. Epub 2011 Nov 14. PMID 22082672